CLINICAL TRIAL: NCT06990282
Title: The Effectiveness of Micro-Needling Technique Using Ozonated Olive Oil on The Treatment of Biofilm Induced Gingivitis & Periodontitis in Comparison to Professional Mechanical Plaque Removal: A Randomized Control Trial.
Brief Title: Micro-Needling Technique Using Ozonated Olive Oil in Periodontal Diseases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Heba Mohammed Hussien Ali, teaching assistant, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNI; fayoum university (Other: educational institution)
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Diseases; Periodontitis and Treatment Need; Gingivitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis | interventions — Percutaneous Collagen Induction; Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: microneedling and ozonated olive oil
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- biofilm induced gingivitis treated with microneedling & topical ozonated olive oil. (Experimental): biofilm induced gingivitis treated with microneedling & topical ozonated olive oil
  Interventions: Other: microneedling; Other: scaling; Biological: Ozonated olive oil
- Periodontitis cases treated by scaling only. (Experimental): Periodontitis cases treated by (PMPR) only.
  Interventions: Other: scaling
- Periodontitis cases treated with microneedling and topical ozonated olive oil. (Experimental): Periodontitis cases treated with microneedle (Dermapen) and topical ozonated olive oil.
  Interventions: Other: microneedling; Other: scaling; Biological: Ozonated olive oil

INTERVENTIONS:
Other: microneedling — gingival microneedling (small holes in gingiva)
  Arms: Periodontitis cases treated with microneedling and topical ozonated olive oil.; biofilm induced gingivitis treated with microneedling & topical ozonated olive oil.
Other: scaling — scaling (plaque removal)
Biological: Ozonated olive oil — ozonated olive oil after microneedling
  Arms: Periodontitis cases treated with microneedling and topical ozonated olive oil.; biofilm induced gingivitis treated with microneedling & topical ozonated olive oil.

SUMMARY:
The research idea is based on using micro-acupuncture therapy with ozone-treated olive oil to improve the condition of patients suffering from gingivitis and periodontitis and comparing it to the scientifically proven conventional treatment. This is a randomized controlled study, and this idea was chosen from the current general trend in medicine, particularly in dentistry, to use natural sources for treatment due to fewer side effects compared to the chemicals used.

DETAILED DESCRIPTION:
The research idea is based on the use of microneedling treatment with ozone-treated olive oil to improve the condition of patients suffering from gingivitis and periodontitis, and to compare this with scientifically proven traditional treatment. It is a randomized controlled study, and this idea has been selected from the general trend currently prevalent in the field of medicine in general and dentistry in particular, which utilizes natural sources for treatment due to the reduced side effects compared to chemical substances used. Research objectives and rationale: to find simple, proven solutions accessible to everyone that rely on natural sources to treat one of the widely spread oral diseases, which negatively affects the patient's overall health and dental health, potentially leading to tooth loss and deteriorating the patient's oral and psychological health as well. The proposed solutions will be compared with scientifically proven solutions that are used regularly to treat this disease. Expected results: that the new intervention using ozone-treated natural olive oil with the microneedling device, which has shown significant effectiveness in various specialties such as dermatology and dentistry, will improve the healing process of the gum membranes And the removal of the inflammations causing deterioration of the membranes surrounding the teeth and the bone resorption around them, which may lead to tooth loss, should improve better than the conventional methods currently used. This involves using laboratory analyses to observe the improvement rates of biological indicators by taking a sample of the gingival crevicular fluid before starting the intervention and afterward, with regular patient follow-up until clinical signs improve. Multiple readings should be taken to assess the improvement in the quality of the membranes, ensuring that the new intervention is simple and accessible to everyone. Operational background: This research is based on numerous previous studies from references, case reports, and analytical studies in the same field published in international scientific journals. Their effectiveness and credibility have been proven by specialists through published systematic reviews, along with the opinions of specialized consultants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Male and female medically free participants
* Patients suffering from biofilm induced gingivitis or periodontitis

Exclusion Criteria:

* Smoking and tobacco related habits
* Non-biofilm induced gingival diseases
* Necrotizing periodontal diseases
* periodontitis as a manifestation of systemic disease
* Third molar tooth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
bleeding on probing | 4 weeks
  Muehlemann & Son index
Plaque index | 4 weeks
  Silness-Loe Plaque Index
probing depth and clinical attachment loss | 4 weeks
  measured in mm using a UNC 15 probe

SECONDARY OUTCOMES:
malondialdehyde and 8-hydroxy-deoxyguanosin level in GCF. | 4 weeks
  measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Nayroz Tarrad, Prof, Study Director — Fayoum University
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: Study Protocol
Time Frame: after publication of the final results
Access Criteria: upon request